CLINICAL TRIAL: NCT07204444
Title: Equipping the Aging Network to Address Social Isolation, Loneliness, and Elevated Suicide Risk Among Vulnerable Older Adults: A Partially Nested Randomized Controlled Trial of the BE WITH Innovation
Brief Title: The BE WITH Project: A Partially Nested Randomized Control Trial (PN-RCT)
Acronym: BE_WITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Georgia State University (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90INNU0021-03-00; 90INNU0021 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-06

CONDITIONS: Older Adults; Mental Health; Depression; Loneliness; Social Isolation; Suicide Ideations; Social Functioning; Quality of Life; Thwarted Belongingness; Perceived Burdensomeness; Help-Seeking Behavior; Suicide Risk
Keywords: mental health clinical trial for older adults
MeSH Terms: conditions — Psychological Well-Being; Depression; Social Isolation; Social Adjustment; Help-Seeking Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Methodologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BE Condition (Experimental): The BE condition which involves receiving treatment from providers trained to foster belongingness and empathy, grounded in the befriending literature (Wiles et al., 2019; Fakoya et al., 2021), and narrative reminiscence (Yousefi, 2015). Aging Network Providers trained in BE provide a "small dose of sincere connection" through 5 core components:
  1. reciprocity: the feeling that both parties are benefiting
  2. intimacy: willingness to share deeply (superficial sharing at first helps build the relationship, but deeper sharing is what leads to positive outcomes)
  3. reliability & respect (calling at the time you say you are going to call creates consistency and reliability, and that the older adult matters
  4. proximity: feeling more connected to people within your community
  5. autonomy: feeling both parties are willingly participating with each connection
  Interventions: Behavioral: standardized and manualized warm calls from providers trained in the BE training
- BE + ASIST Condition (Experimental): The BE + ASIST condition includes the BE training + the aging variant of LivingWorks ASIST (Applied Suicide Intervention Skills Training; Lang et al., 2013). Analogous to CPR, paraprofessionals can learn "suicide first aid." Providers trained in ASIST are equipped to do a 6 step model (Pathway for Assisting Life (PAL)) to help stabilize a person at risk of suicide at the moment it needed the most. The PAL model matches six needs of the older adult-at-risk with six tasks of the treatment provider. These include (1) exploring invitations (i.e. voluntary stopping of eating and drinking, withholding medical treatment, etc.), 2. asking directly about suicide, 3. sincerely hearing the story about suicide, 4. working effectively with ambivalence about dying, and offering a 3rd option (to stay safe for now), 5. developing a mutually endorsed safety plan, and 6. confirming actions (asking the older adult to repeat the plan back to the provider)
  Interventions: Behavioral: standardized and manualized warm calls from providers trained in the BE training + ASIST training
- Control (No Intervention): participants randomized to this condition will not receive call dosages during the clinical trial. However, they will have the option to receive call dosages after the 8 weeks have concluded.

INTERVENTIONS:
Behavioral: standardized and manualized warm calls from providers trained in the BE training — Weekly call dosages averaging 20-30 minutes each, for 8 weeks duration
  Arms: BE Condition
Behavioral: standardized and manualized warm calls from providers trained in the BE training + ASIST training — Weekly call dosages averaging 20-30 minutes each, for 8 weeks duration
  Arms: BE + ASIST Condition

SUMMARY:
The goal of this clinical trial is to learn if the BE WITH (Belonging through Empathy With Intentional Targeted Helping) innovation delivered to older adults improves their mental health. It will also learn about the treatment components that led to improvements. The main questions it aims to answer are:

1. Over the course of the 8 week standardized and manualized warm calling treatment, are mental health outcomes improved for the BE and BE + ASIST (Applied Suicide Intervention Skills Training) treatment conditions relative to a control group?
2. Are there differential outcomes for older adults who start the treatment at low, medium, or high risk? (as defined by a baseline aggregate of measures)?
3. How is this improvement manifested for particular aspects of mental health (i.e. depression, social needs, suicide desire, and overall quality of life)?

Participants will:

1. answer questions from a trained data collector to get their baseline,
2. receive 8 weeks of warm calls for 2 months (if assigned to one of the 2 treatment conditions, if assigned to control they will have the option to receive treatment at a later time), and (c) be assessed every 2 weeks.

DETAILED DESCRIPTION:
This study is a partially nested randomized controlled trial research design (PN-RCT) with a two-level structure of clients (level-1) nested within callers (level-2) for the two treatment conditions which receive calls. Given that outcomes for older adults receiving calls from the same treatment provider may be more similar than for those who receive calls from a different provider, the use of multilevel modeling can account for these data dependencies. The investigators will be investigating 1) how our BE WITH (Belonging through Empathy With Intentional Targeted Helping) innovation reduces social isolation, loneliness, and elevated suicidality among home delivered meal and former congregate meal clients and improves their social support and well-being. Social isolation, loneliness, and elevated suicidality will be operationalized through a combination of validated psychometric measures taken before, during, and after the structured 8-week intervention. For older adults receiving calls, data from validated measures will be triangulated with behavioral observations of the older adults' emotional states based upon a structured analysis of recorded audio files. The investigators hypothesize that older adults in both treatment conditions will have reduced: social isolation, loneliness, depression, mental health distress, and suicide desire; and they will have increased: social connection, social support, and well-being over time and in comparison to those in the control condition. The investigators will also investigate 2) how BE WITH improves the frequency of empathic and suicide intervention best practice behaviors by trained nutrition service providers. This will be demonstrated in both real-world settings and in situations where a research confederate presents a clinically heightened risk of social isolation, loneliness, and elevated suicidality. Evaluation of counseling skills and suicide intervention skills is challenging, as observations of caregivers working with clients are required. We hypothesize that those trained in both conditions will demonstrate positive global counseling behaviors; however, those trained in BE WITH will more often employ suicide intervention practices when needed.

ELIGIBILITY:
Inclusion Criteria for older adult participants:

1. Provision of verbal informed consent,
2. Classify as an Older Adult (55+),
3. Stated willingness and ability to comply with all study procedures,
4. Receive nutrition services through the Aging Services Network (i.e. either HDM (home delivered meals services) or CM (congregate meals)), and
5. Be affiliated with one of the 25 senior centers we will contract with through a Memorandum of Understanding.

Inclusion Criteria for trained providers:

1. Provision of written informed consent,
2. State willingness to comply with all study procedures,
3. Be a staff or volunteer within the ASN (Aging Services Network), specifically within the 25 senior centers we are working with,
4. Meet criteria identified by Wymann and colleagues (2009) for being a "natural helpers" (i.e. be warm, empathic, and having ongoing interaction with participants through one's job role), and
5. Be recommended by the senior center leadership as meeting these qualifications.

Exclusion Criteria for older adult participants:

1. Had a dementia diagnosis, or another form of cognitive impairment, and/or hearing impairment that would preclude phone conversation, and
2. Participation in another warm calling behavioral treatment or intervention study simultaneously occurring in this state.

The reasons given to exclude participants with dementia/cognitive impairment diagnoses from large-scale clinical research are partially related to the concern of a potential risk of abuse and exploitation. Further, those with cognitive impairment are not able to give informed consent, and there are measurement challenges with behavioral health data.

Exclusion Criteria for trained helpers:

1. Does not have ongoing interactions with potential old adult participants (i.e. is a part of an optimized nutrition service provider in which they do not serve the same older adults consistently over time), and
2. Participation in another warm calling behavioral treatment or intervention study simultaneously occurring in this state.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura R Shannonhouse, PhD, Principal Investigator — University of Florida
Locations (1):
- Older Adults' Homes; Treatment Provided Over the Phone, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant data for several reasons:
  1. Ensuring participant privacy: De-identification and secure data management are crucial to protect participant information,
  2. Financial resources: Data sharing requires additional resources for data preparation, data sharing agreements, storage, and management which were not included in this grant,
  3. Addressing potential biases: Sharing data must be done in a way that minimizes bias and allows for fair and transparent use.

REFERENCES:
- [Background] Hill, C. E., Knox, S., Thompson, B.J., & Williams, E. N., (1997). A guide to conducting consensual qualitative research. The Counseling Psychologist, 25, 517-572. 44Hill, C. E., Knox, S., Thompson, B. J., Williams, E. N., Hess, S. A., & Ladany, N. (2005). Consensual qualitative research: An update. Journal of Counseling Psychology, 52, 196-205.
- [Background] Efron, B. (1971). Forcing a sequential experiment to be balanced. Biometrika, 58(3), 403-417.
- [Background] Lang, W. A., Ramsay, R. F., Tanney, B. L., Kinzel, T., Turley, B., & Tierney, R. J. (2013). ASIST trainer manual ( 11th ed.). Calgary, Alberta, Canada: LivingWorks Education.
- [Background] Caplan, G. (1964). Principles of preventive psychiatry.
- [Background] Yousefi Z, Sharifi K, Tagharrobi Z, Akbari H. The Effect of Narrative Reminiscence on Happiness of Elderly Women. Iran Red Crescent Med J. 2015 Nov 7;17(11):e19612. doi: 10.5812/ircmj.19612. eCollection 2015 Nov. PMID 26734470
- [Background] Fakoya OA, McCorry NK, Donnelly M. How do befriending interventions alleviate loneliness and social isolation among older people? A realist evaluation study. PLoS One. 2021 Sep 9;16(9):e0256900. doi: 10.1371/journal.pone.0256900. eCollection 2021. PMID 34499682
- [Background] Dale M, Fortin MJ. Spatial analysis: a guide for ecologists. Cambridge University Press; 2014.
- [Background] Tseng C, Shao Y. Sample size growth with an increasing number of comparisons. J Probab Stat. 2012;2012:1-10.
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Background] Chow SC, Shao J, Wang H, Lokhnygina Y. Sample size calculations in clinical research. Chapman and Hall; 2017.
- [Background] Lohr S, Schochet PZ, Sanders E. Partially Nested Randomized Controlled Trials in Education Research: A Guide to Design and Analysis. NCER 2014-2000. National Center for Education Research; 2014.
- [Background] Friedman LM, Furberg CD, DeMets DL, Reboussin DM, Granger CB. Fundamentals of clinical trials. Springer; 2015.
- [Background] Piantadosi S. Clinical trials: a methodologic perspective. John Wiley & Sons; 2017.
- [Background] Mabli J, Gearan E, Cohen R, Niland K, Redel N, Panzarella E, Carlson B. Evaluation of the effect of the Older Americans Act Title III-C Nutrition Services Program on participants' food security, socialization, and diet quality. Washington, DC: US Department of Health and Human Services, Administration for Community Living; April 1, 2017-07. Retrieved from https://www.sustaintool.org/psat/.
- [Background] Mabli J, Redel N, Cohen R, Panzarella E, Hu M, Carlson B. Process evaluation of Older Americans Act Title III-C nutrition services program. Washington, DC: US Department of Health and Human Services, Administration for Community Living; 2017-02
- [Background] Wright L, Vance L, Sudduth C, Epps JB. The Impact of a Home-Delivered Meal Program on Nutritional Risk, Dietary Intake, Food Security, Loneliness, and Social Well-Being. J Nutr Gerontol Geriatr. 2015;34(2):218-27. doi: 10.1080/21551197.2015.1022681. PMID 26106989
- [Background] Sparling TM, Cheng B, Deeney M, Santoso MV, Pfeiffer E, Emerson JA, Amadi FM, Mitu K, Corvalan C, Verdeli H, Araya R, Kadiyala S. Global Mental Health and Nutrition: Moving Toward a Convergent Research Agenda. Front Public Health. 2021 Oct 8;9:722290. doi: 10.3389/fpubh.2021.722290. eCollection 2021. PMID 34722437
- [Background] 2020 Global Nutrition Report. Action on equity to end malnutrition. Bristol, UK: Development Initiatives. Retrieved from https://globalnutritionreport.org/documents/566/2020_Global_Nutrition_Report_2hrssKo.pdf.
- [Background] Lobato ZM, Almeida da Silva AC, Lima Ribeiro SM, Biella MM, Santos Silva Siqueira A, Correa de Toledo Ferraz Alves T, Machado-Vieira R, Borges MK, Oude Voshaar RC, Aprahamian I. Nutritional Status and Adverse Outcomes in Older Depressed Inpatients: A Prospective Study. J Nutr Health Aging. 2021;25(7):889-894. doi: 10.1007/s12603-021-1638-y. PMID 34409967
- [Background] Fullen MC, Lawson GF, Sharma J. Analyzing the impact of the Medicare coverage gap on counseling professionals: Results of a national study. J Couns Dev. 2020;98:207-19.
- [Background] Perissinotto CM, Stijacic Cenzer I, Covinsky KE. Loneliness in older persons: a predictor of functional decline and death. Arch Intern Med. 2012 Jul 23;172(14):1078-83. doi: 10.1001/archinternmed.2012.1993. PMID 22710744
- [Background] Meals on Wheels America. More Than A Meal Pilot Research Study. https://www.mealsonwheelsamerica.org/learn-more/research/more-than-a-meal/pilotresearch-study. 2015.
- [Result] Shannonhouse L, Lin YD, Shaw K, Wanna R, Porter M. Suicide intervention training for college staff: Program evaluation and intervention skill measurement. J Am Coll Health. 2017 Oct;65(7):450-456. doi: 10.1080/07448481.2017.1341893. Epub 2017 Jun 19. PMID 28628372
- [Result] Wyman PA, Brown CH, Inman J, Cross W, Schmeelk-Cone K, Guo J, Pena JB. Randomized trial of a gatekeeper program for suicide prevention: 1-year impact on secondary school staff. J Consult Clin Psychol. 2008 Feb;76(1):104-15. doi: 10.1037/0022-006X.76.1.104. PMID 18229988
- [Result] Witte TK, Merrill KA, Stellrecht NE, Bernert RA, Hollar DL, Schatschneider C, Joiner TE Jr. "Impulsive" youth suicide attempters are not necessarily all that impulsive. J Affect Disord. 2008 Apr;107(1-3):107-16. doi: 10.1016/j.jad.2007.08.010. Epub 2007 Sep 4. PMID 17804082
- [Result] Van Orden KA, Witte TK, Cukrowicz KC, Braithwaite SR, Selby EA, Joiner TE Jr. The interpersonal theory of suicide. Psychol Rev. 2010 Apr;117(2):575-600. doi: 10.1037/a0018697. PMID 20438238
- [Result] Fullen MC, Smith JL, Clarke PB, Westcott JB, McCoy R, Tomlin CC. Holistic Wellness Coaching for Older Adults: Preliminary Evidence for a Novel Wellness Intervention in Senior Living Communities. J Appl Gerontol. 2023 Mar;42(3):427-437. doi: 10.1177/07334648221135582. Epub 2022 Oct 28. PMID 36307916
- [Result] Middleton G, Patterson KA, Muir-Cochrane E, Velardo S, McCorry F, Coveney J. The Health and Well-being Impacts of Community Shared Meal Programs for Older Populations: A Scoping Review. Innov Aging. 2022 Oct 27;6(7):igac068. doi: 10.1093/geroni/igac068. eCollection 2022. PMID 36588625
- [Result] Porter Starr K, Fischer JG, Johnson MA. Eating behaviors, mental health, and food intake are associated with obesity in older congregate meal participants. J Nutr Gerontol Geriatr. 2014;33(4):340-56. doi: 10.1080/21551197.2014.965375. PMID 25424510
- [Result] Fullen MC, Shannonhouse LR, Mize MC, Miskis C. Mental health distress in homebound older adults: Importance of the aging network. Aging Ment Health. 2021 Aug;25(8):1580-1584. doi: 10.1080/13607863.2020.1758920. Epub 2020 Apr 29. PMID 32347109
- [Result] Grajek M, Krupa-Kotara K, Bialek-Dratwa A, Sobczyk K, Grot M, Kowalski O, Staskiewicz W. Nutrition and mental health: A review of current knowledge about the impact of diet on mental health. Front Nutr. 2022 Aug 22;9:943998. doi: 10.3389/fnut.2022.943998. eCollection 2022. PMID 36071944
- [Result] Walton K, do Rosario VA, Pettingill H, Cassimatis E, Charlton K. The impact of home-delivered meal services on the nutritional intake of community living older adults: a systematic literature review. J Hum Nutr Diet. 2020 Feb;33(1):38-47. doi: 10.1111/jhn.12690. Epub 2019 Jul 2. PMID 31266095
- [Result] Thomas KS, Smego R, Akobundu U, Dosa D. Characteristics of Older Adults on Waiting Lists for Meals on Wheels: Identifying Areas for Intervention. J Appl Gerontol. 2017 Oct;36(10):1228-1242. doi: 10.1177/0733464815614918. Epub 2015 Nov 23. PMID 26597791
- [Result] Van Orden K, Conwell Y. Suicides in late life. Curr Psychiatry Rep. 2011 Jun;13(3):234-41. doi: 10.1007/s11920-011-0193-3. PMID 21369952
- [Result] Boulos C, Salameh P, Barberger-Gateau P. Social isolation and risk for malnutrition among older people. Geriatr Gerontol Int. 2017 Feb;17(2):286-294. doi: 10.1111/ggi.12711. Epub 2016 Jan 21. PMID 26790629
- [Result] Azizi-Zeinalhajlou A, Mirghafourvand M, Nadrian H, Samei Sis S, Matlabi H. The contribution of social isolation and loneliness to sleep disturbances among older adults: a systematic review. Sleep Biol Rhythms. 2022 Feb 28;20(2):153-163. doi: 10.1007/s41105-022-00380-x. eCollection 2022 Apr. PMID 38469248
- [Result] Shankar A, McMunn A, Banks J, Steptoe A. Loneliness, social isolation, and behavioral and biological health indicators in older adults. Health Psychol. 2011 Jul;30(4):377-85. doi: 10.1037/a0022826. PMID 21534675
- [Result] Taylor HO. Social Isolation's Influence on Loneliness among Older Adults. Clin Soc Work J. 2020 Mar;48(1):140-151. doi: 10.1007/s10615-019-00737-9. Epub 2019 Dec 23. PMID 33343042
- [Result] Nicholson NR. A review of social isolation: an important but underassessed condition in older adults. J Prim Prev. 2012 Jun;33(2-3):137-52. doi: 10.1007/s10935-012-0271-2. PMID 22766606
- [Result] Coyle CE, Dugan E. Social isolation, loneliness and health among older adults. J Aging Health. 2012 Dec;24(8):1346-63. doi: 10.1177/0898264312460275. Epub 2012 Sep 23. PMID 23006425
- [Result] Finlay JM, Kobayashi LC. Social isolation and loneliness in later life: A parallel convergent mixed-methods case study of older adults and their residential contexts in the Minneapolis metropolitan area, USA. Soc Sci Med. 2018 Jul;208:25-33. doi: 10.1016/j.socscimed.2018.05.010. Epub 2018 May 4. PMID 29758475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in the study; Trained Providers/Helpers were not considered enrolled
Groups:
- BE Condition: The BE condition which involves receiving treatment from providers trained to foster belongingness and empathy, grounded in the befriending literature (Wiles et al., 2019; Fakoya et al., 2021), and narrative reminiscence (Yousefi, 2015). Aging Network Providers trained in BE provide a "small dose of sincere connection" through 5 core components:
  1. reciprocity: the feeling that both parties are benefiting
  2. intimacy: willingness to share deeply (superficial sharing at first helps build the relationship, but deeper sharing is what leads to positive outcomes)
  3. reliability & respect (calling at the time you say you are going to call creates consistency and reliability, and that the older adult matters
  4. proximity: feeling more connected to people within your community
  5. autonomy: feeling both parties are willingly participating with each connection
  standardized and manualized warm calls from providers trained in the BE training: Weekly call dosages averaging 20-30 minutes each, for 8 weeks duration
Period: Overall Study
Arm/Group | BE Condition | BE + ASIST Condition | Control
Started | 236 | 227 | 208
Completed | 183 | 176 | 179
Not Completed | 53 | 51 | 29
Not completed — Medical/Hospitalization | 6 | 9 | 6
Not completed — Treatment Provider Issue | 1 | 3 | 0
Not completed — Withdrawal by Subject | 11 | 5 | 5
Not completed — Death | 3 | 6 | 1
Not completed — Unable To Reach | 29 | 26 | 17
Not completed — Protocol Deviation | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BE Condition | BE + ASIST Condition | Control | Total
Number analyzed (Participants) | 236 | 227 | 208 | 671
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing record for age for three individuals
  years
    number analyzed (Participants) | 235 | 225 | 208 | 668
    (all) | 73.74 (8.60) | 73.97 (8.54) | 73.75 (8.70) | 73.82 (8.60)
Age, Customized [Count of Participants; unit: Participants]
  Not Reported | 1 | 2 | 0 | 3
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 25 | 23 | 76
  >=65 years | 207 | 200 | 185 | 592
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 150 | 149 | 126 | 425
  Male | 86 | 77 | 82 | 245
  Transgender, Male to Female | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 3 | 11
  Not Hispanic or Latino | 230 | 223 | 205 | 658
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3 | 6
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 132 | 129 | 129 | 390
  White | 88 | 83 | 64 | 235
  More than one race | 7 | 5 | 9 | 21
  Unknown or Not Reported | 8 | 8 | 2 | 18
Region of Enrollment [Number; unit: participants]
  United States | 236 | 227 | 208 | 671

OUTCOME MEASURES:

1. Primary Outcome: Social Provisions Scale (SPS-5)
Description: The Social Provisions Scale (SPS-5) is a 5-item measure used to evaluate a participant's level of social support. It is a shortened version of the 10-item SPS and designed for use in research studies to reduce participant burden while maintaining strong psychometric properties. The SPS is based on a theory of social support developed by Irwin Weiss and uses one positive item to assess the social provisions of Attachment, Guidance, Social Integration, Reliable alliance, and Reassurance of worth. Each item is rated on a 4-point Likert scale, from "Strongly Disagree" to "Strongly Agree". Sample items include, "There is someone I could talk to about important decisions in my life", "I feel part of a group of people who share my attitudes and beliefs", and "There are people I can count on in an emergency." A total score is calculated by summing the responses to the 5 questions. The scores can range from 5 to 20, with higher scores indicating higher levels of perceived social support.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: Not all individuals completed every survey question. As a result, the total number of responses for each survey was less than or equal to the arm size.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition | Control
Number analyzed (Participants) | 236 | 227 | 208
score on a scale
  Baseline: number analyzed (Participants) | 236 | 225 | 208
  Baseline | 16.88 (3.423) | 17 (3.328) | 17.16 (3.047)
  Week 2: number analyzed (Participants) | 195 | 188 | 195
  Week 2 | 17.34 (3.191) | 17.51 (2.820) | 16.98 (3.095)
  Week 4: number analyzed (Participants) | 184 | 182 | 186
  Week 4 | 17.22 (3.366) | 17.54 (2.974) | 17.03 (3.100)
  Week 6: number analyzed (Participants) | 172 | 172 | 182
  Week 6 | 17.19 (3.148) | 17.35 (3.037) | 17.21 (3.164)
  Week 8: number analyzed (Participants) | 181 | 176 | 179
  Week 8 | 17.60 (3.428) | 17.78 (2.868) | 17.18 (3.112)

2. Primary Outcome: University of California, Los Angeles Loneliness Scale
Description: The three-item UCLA Loneliness Scale (Hughes et al., 2004) is a widely used instrument for measuring subjective feelings of loneliness. The scale assesses three core dimensions of loneliness through corresponding items: relational connectedness ("How often do you feel that you lack companionship?"), social connectedness ("How often do you feel left out?"), and self-perceived isolation ("How often do you feel isolated from others?"). Participants respond using a 3-point scale ranging from "hardly ever" to "often." Total scores range from 3 to 9, with higher scores indicating greater loneliness. The scale demonstrates good psychometric properties in middle-aged and older adult populations.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition | Control
Number analyzed (Participants) | 236 | 227 | 208
score on a scale
  Baseline | 5.131 (2.016) | 5.035 (1.984) | 4.697 (1.849)
  Week 2: number analyzed (Participants) | 196 | 188 | 195
  Week 2 | 4.786 (1.923) | 4.702 (1.829) | 4.846 (1.761)
  Week 4: number analyzed (Participants) | 184 | 182 | 186
  Week 4 | 4.614 (1.807) | 4.670 (1.854) | 4.737 (1.795)
  Week 6: number analyzed (Participants) | 172 | 172 | 183
  Week 6 | 4.628 (1.880) | 4.372 (1.761) | 4.525 (1.800)
  Week 8: number analyzed (Participants) | 181 | 176 | 179
  Week 8 | 4.448 (1.717) | 4.455 (1.703) | 4.346 (1.771)

3. Primary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: The GAD-7 is a 7-item questionnaire designed to assess the symptoms of Generalized Anxiety Disorder (GAD). Each item describes a common GAD symptom and is rated on a four-point scale (0-3) based on how often the individual has experienced that symptom over the past 2 weeks. The 7 questions assess feelings such as nervousness, inability to control worrying, trouble relaxing, restlessness, irritability, and feeling afraid. Sample items include, "how often have you felt nervous, anxious, or on edge", "how often have you worried too much about different things", "how often have you had trouble relaxing", and "fFelt afraid as if something awful might happen." Total scores range from 0 to 21, with higher scores indicating increased anxiety severity. Scores are categorized as: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety).
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition | Control
Number analyzed (Participants) | 236 | 227 | 208
score on a scale
  Baseline: number analyzed (Participants) | 236 | 226 | 208
  Baseline | 4.919 (5.447) | 4.544 (5.135) | 4.433 (4.838)
  Week 2: number analyzed (Participants) | 195 | 188 | 195
  Week 2 | 4.005 (4.713) | 4.074 (5.019) | 4.851 (4.778)
  Week 4: number analyzed (Participants) | 184 | 181 | 186
  Week 4 | 4.277 (5.103) | 4.083 (4.893) | 4.489 (4.542)
  Week 6: number analyzed (Participants) | 172 | 172 | 183
  Week 6 | 3.628 (4.318) | 3.616 (4.928) | 4.295 (5.025)
  Week 8: number analyzed (Participants) | 180 | 174 | 179
  Week 8 | 3.794 (4.759) | 3.546 (4.586) | 3.855 (4.670)

4. Primary Outcome: Patient Health Questionnaire - PHQ-9
Description: The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure to assess depressive symptoms in the past 2 weeks (Kroenke et al., 2001). The scale items correspond to the 9 diagnostic criteria for major depressive disorder. Respondents rate the frequency of each symptom on a 4-point scale ranging from "not at all" to "nearly every day." Sample items include "Little interest or pleasure in doing things" and "Poor appetite or overeating." Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. The PHQ-9 includes an additional functional impairment item that assesses how much the problems have affected the respondents' daily activities. The scale has shown strong psychometric properties across diverse populations. Among U.S. older adults, the PHQ-9 showed high sensitivity (88%) and specificity (80%) for identifying major depression, as well as the combination of major and minor depression (Phelan et al., 2010).
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition | Control
Number analyzed (Participants) | 236 | 227 | 208
score on a scale
  Baseline: number analyzed (Participants) | 203 | 188 | 171
  Baseline | 5.768 (5.655) | 5.404 (5.419) | 5.433 (5.318)
  Week 2: number analyzed (Participants) | 195 | 187 | 187
  Week 2 | 5.077 (5.641) | 4.759 (4.742) | 5.342 (4.860)
  Week 4: number analyzed (Participants) | 184 | 182 | 186
  Week 4 | 4.908 (5.709) | 4.692 (5.287) | 5.349 (5.134)
  Week 6: number analyzed (Participants) | 172 | 172 | 183
  Week 6 | 4.680 (5.314) | 3.797 (4.263) | 5.098 (5.467)
  Week 8: number analyzed (Participants) | 180 | 175 | 178
  Week 8 | 4.661 (5.275) | 4.229 (4.901) | 5.017 (5.431)

5. Primary Outcome: Short Form Health Survey (SF-12)
Description: The Short Form Health Survey (SF-12) is a self-reported outcome measure to assess health-related quality of life. The raw answers from the 12 questions are processed to produce two main, standardized summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). We only used the MCS factor in this study as the treatment is targeting mental health. The MCS computed score has a range from 17 to 64 in the analysis and was based on the linear combination of six computed, generated, iterated weights. A low Mental Component Summary (MCS) score indicates poorer self-perceived mental health and lower health-related quality of life.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition | Control
Number analyzed (Participants) | 236 | 227 | 208
score on a scale
  Baseline | 44.02 (11.61) | 44.17 (11.61) | 44.24 (11.78)
  Week 2: number analyzed (Participants) | 196 | 188 | 195
  Week 2 | 45.59 (11.57) | 45.56 (11.30) | 44.73 (10.71)
  Week 4: number analyzed (Participants) | 184 | 182 | 186
  Week 4 | 46.79 (12.19) | 46.42 (11.37) | 45.32 (11.07)
  Week 6: number analyzed (Participants) | 172 | 171 | 183
  Week 6 | 46.49 (11.86) | 47.46 (10.85) | 45.59 (11.24)
  Week 8: number analyzed (Participants) | 181 | 176 | 178
  Week 8 | 47.19 (11.89) | 47.52 (11.48) | 46.07 (10.93)

6. Primary Outcome: Interpersonal Needs Questionnaire (INQ-15)
Description: The Interpersonal Needs Questionnaire (INQ; Van Orden et al., 2012) was used to evaluate thwarted belongingness and perceived burdensomeness through 15 items. We used an adapted version tailored specifically for older adults which includes 3-point Likert scale ranging from 1 (Not at all true for me) to 3 (Very true for me). The instrument includes 2 sets of characteristics: (1) the 9-item Thwarted Belongingness (e.g., "I feel disconnected from other people."); and (2) the 6-item Perceived Burdensomeness (e.g., "I think my death would be a relief to the people in my life."). Six questions from the Thwarted Belongingness subscale were reverse-coded when the overall score across questions was computed due to the nature of those questions. In particular, the total score on the INQ is calculated by summing the questions responses to all items and reversing the appropriate ones. As a result, greater scores on each subscale reflect higher levels of the respective construct being measured.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition | Control
Number analyzed (Participants) | 236 | 227 | 208
score on a scale
  Baseline: number analyzed (Participants) | 232 | 224 | 202
  Baseline | 19.06 (5.396) | 18.83 (5.336) | 18.59 (4.742)
  Week 2: number analyzed (Participants) | 195 | 188 | 194
  Week 2 | 18.68 (5.384) | 18.36 (5.028) | 18.24 (4.497)
  Week 4: number analyzed (Participants) | 184 | 182 | 184
  Week 4 | 18.35 (5.341) | 18.05 (5.113) | 18.36 (5.137)
  Week 6: number analyzed (Participants) | 172 | 172 | 181
  Week 6 | 18.77 (5.163) | 17.81 (4.757) | 18.15 (5.353)
  Week 8: number analyzed (Participants) | 180 | 174 | 174
  Week 8 | 18.22 (5.062) | 17.89 (5.253) | 18.05 (4.982)

7. Secondary Outcome: Session Rating Scale
Description: The 4-item Session Rating Scale is a therapeutic practice measure that treatment recipients complete after receiving treatment. This allows trained helpers to make real-time adjustments to improve treatment effectiveness and prevent dropout. Participants marked their responses on a Likert-Scale, ranging from 0 to 10, representing: (a) the quality of the therapeutic relationship, (b) agreement on goals and topics, (c) the relevance and fit of the treatment provider's approach, and (d) the overall effectiveness of the treatment dosage. The scores for each domain were summed to generate a total possible score of 40. A total score below 36 or a score below 9 on any single item is a potential indicator of concern, which should prompt the therapist to discuss the issue openly with the client and make necessary adjustments to the session's direction or approach.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 8
Population: The SRS is designed to provide therapists with immediate feedback on how the client is experiencing the therapeutic relationship and session. The study control group does not applicable for this measurement. Nothing is measured at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BE Condition | BE + ASIST Condition
Number analyzed (Participants) | 236 | 227
score on a scale
  Week 2: number analyzed (Participants) | 194 | 187
  Week 2 | 38.65 (3.809) | 38.34 (3.186)
  Week 4: number analyzed (Participants) | 183 | 181
  Week 4 | 38.86 (3.106) | 38.86 (3.227)
  Week 6: number analyzed (Participants) | 172 | 172
  Week 6 | 38.92 (2.652) | 38.89 (3.010)
  Week 8: number analyzed (Participants) | 179 | 174
  Week 8 | 39.28 (2.198) | 39.24 (2.688)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from subject consent up to 200 days.
Arm/Group | BE Condition | BE + ASIST Condition | Control
All-Cause Mortality (participants affected / at risk) | 3/236 | 6/227 | 1/208
Serious Adverse Events (participants affected / at risk) | 6/236 | 9/227 | 6/208
Other Adverse Events (participants affected / at risk) | 0/236 | 0/227 | 0/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BE Condition (N=236) | BE + ASIST Condition (N=227) | Control (N=208)
Medical/Hospitalization (General disorders) | 6 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT07204444/Prot_SAP_000.pdf